CLINICAL TRIAL: NCT04130100
Title: To Evaluate the Safety and Efficacy of Dental Pulp Mesenchymal Stem Cells in the Treatment of Primary Mild to Moderate Knee Osteoarthritis Using Sodium Hyaluronate as a Parallel Control.
Brief Title: Clinical Study of Pulp Mesenchymal Stem Cells in the Treatment of Primary Mild to Moderate Knee Osteoarthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAR-T (Shanghai) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT005SH002
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: low dose of dental pulp mesenchymal stem cells high dose of dental pulp mesenchymal stem cells Sodium hyaluronate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose of Mesenchymal stem cell (Experimental): Patients receiving intraarticular injection of low dose of mesenchymal stem cells.
  Interventions: Biological: Low Dose of Mesenchymal stem cell
- High Dose of Mesenchymal stem cell (Experimental): Patients receiving intraarticular injection of high dose of mesenchymal stem cells.
  Interventions: Biological: High Dose of Mesenchymal stem cell
- Sodium Hyaluronate (Active Comparator): Patients receiving intraarticular injection of Sodium Hyaluronate
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Biological: Low Dose of Mesenchymal stem cell — Mesenchymal stem cell injection
  Other Names: 1
  Arms: Low Dose of Mesenchymal stem cell
Biological: High Dose of Mesenchymal stem cell — Mesenchymal stem cell injection
  Other Names: 2
  Arms: High Dose of Mesenchymal stem cell
Drug: Sodium Hyaluronate — Sodium Hyaluronate injection
  Other Names: 3
  Arms: Sodium Hyaluronate

SUMMARY:
To evaluate the clinical efficacy and safety of dental pulp mesenchymal stem cells in the treatment of primary mild to moderate knee osteoarthritis through a comparative study with sodium hyaluronate.

20 participants will receive low dose of dental pulp mesenchymal stem cells, 20 participants will receive high dose and another 20 participants will receive sodium hyaluronate

DETAILED DESCRIPTION:
60 participants will receive to evaluate the clinical efficacy and safety of dental pulp mesenchymal stem cells in the treatment of primary mild to moderate knee osteoarthritis through a comparative study with sodium hyaluronate and verify the basis of dental pulp mesenchymal stem cells in the treatment of primary knee osteoarthritis, and to explore a more effective and safe clinical treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Complying with the diagnostic criteria for primary knee osteoarthritis revised by the American Rheumatological Association (1995), age 40-70 years, gender-free.
2. For patients with mild to moderate knee arthritis, the WOMAC score of knee joint was less than 120.
3. X-ray Kellgren-Lawrence was used to evaluate the grade I, II and III of osteoarthritis.
4. Fertility patients should take effective contraceptive measures until the end of follow-up. Fertility women should exclude the possibility of early pregnancy, that is, HCG negative test in early pregnancy.
5. Voluntary participation in this clinical study, can cooperate with doctors to carry out research, stop all medical measures for knee arthritis for more than 2 weeks, and sign the informed consent of patients.

Exclusion Criteria:

(1) Those with other diseases that may affect the knee joint, such as rheumatoid arthritis, ankylosing spondylitis, rheumatoid arthritis, gout and other rheumatic diseases, bone tumors, osteoporosis, bone tuberculosis or obvious history of acute trauma, resulting in meniscus injury, ligament rupture and vascular nerve injury; those with previous history of femur, tibial plateau, tibia and fibula fracture. The patients with gonarthritis, the patients with knee joint and surrounding skin infection were not cured.

2) Patients who have undergone surgery and other factors affecting the efficacy of the treatment. Patients with severe deformities or even deformities of the knee joint, who need surgical treatment. Patients who have received knee joint irrigation or arthroscopic examination within one year.

3) Patients with systemic cancer tendency or cancer and patients with systemic infection in active stage.

4) Patients with severe heart, lung, liver, kidney, blood system, endocrine system and immune deficiency, or abnormal laboratory biochemical indicators, namely: hemoglobin (Hb) < 9 g/dL, white blood cell (WBC) > 15 x 109/L, platelet (Pt) < 100 x 109/L, glutamic oxalate transaminase (AST) and alanine aminotransferase (ALT) > 1.5 times normal upper limit; serum creatinine > 1.5 times normal upper limit.

5) Physical history or clinical manifestations with bleeding tendency, including patients currently using anticoagulants.

6) Patients with uncontrollable epileptic seizures, psychosis or Alzheimer's disease who are unable to complete the scale.

7) Pregnant or lactating women, legal disabled patients (blind, deaf, dumb, mentally retarded, physically disabled), drug addiction and other adverse drug addiction.

8) Patients with contraindications or allergies were examined and treated in this study.

9) Those who have participated in other clinical studies within one month.

10) Researchers consider it inappropriate for patients to participate in this clinical study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Kellgren and Lawrence's rating | 12 month
  X-ray imaging was used to evaluate the degree of improvement in knee joint structure
WOMAC score | 12 month
  WOMAC score decreased

SECONDARY OUTCOMES:
Volume of femoral surface of knee joint on MRI | 12 month
  Changes of volume of lateral femoral condylar, medial femoral condylar, lateral tibial condylar, medial tibial condylar and posterior patellar articular surfaces on MRI
relaxation time of femoral surface of knee joint on MRI | 12 month
  Changes of relaxation time (T1 condylar, T2 condylar, T2*) of lateral femoral condylar, medial femoral condylar, lateral tibial condylar, medial tibial condylar and posterior patellar articular surfaces on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Dongbao Zhao, Doctor, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No